CLINICAL TRIAL: NCT06416683
Title: Study of the Atezolizumab and Bevacizumab Combination Recommended in a Multidisciplinary Consultation Meeting in Caen for Hepatocellular Carcinoma.
Brief Title: Atezolizumab and Bevacizumab Combination Recommended in a Multidisciplinary Consultation Meeting in Caen for Hepatocellular Carcinoma (ABCHCaen)
Acronym: ABCHCaen
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: ABCHCaen
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-05

CONDITIONS: Atezolizumab and Bevacizumab in Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In France primary liver cancers (PLC) is the fourth leading cause of cancer-related death in men, and the seventh in women. The number of new cases per year is predicted to increase by 26.5% between 2020 and 2040. Hepatocellular carcinoma (HCC) account for 75% to 85% of PLC. It occurs mostly on cirrhotic livers. Diagnosis remains late in almost half of the patients so that a palliatif treatment is frequent. In advanced cases sorafenib has been so far the first line systemic therapy since 2008. In 2020 a phase 3 study has demonstrated a better overall survival in patients treated with bevacizumab associated with atezolizumab as compared to sorafenib (19.2 months vs 13.4 months) and a better quality of life. Noweday immunotherapy is recommended in first line in cases of ECOG 0/1 unresectable HCC without liver insufficiency. However the study included 70% of viral liver diseases while HCC are related to alcohol and steatohepatitis in 50% of cases in France. Moreover patients with high risk of oesophageal variceal bleeding were excluded. Recent real life data published worldwide confirm the bitherapy efficacy and good tolerability. By contrast french data are scarces, with a single serie of 43 patients in which median overall survival was estimated to 12 months. Our main aim is to determine the overall survival of HCC patients treated with atezolizumab and bevacizumab in Caen from april 2021.

ELIGIBILITY:
Inclusion Criteria:

* age superior or equal to 18 years
* patients with advanced hepatocellular carcinoma
* treatment validated in multidisciplinary consultation meeting

Exclusion Criteria:

* patients with another kind of liver cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with advanced hepatocellular carcinoma whose treatment with Atezolizumab and Bevacizumab has been validated in a multidisciplinary consultation meeting
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years
  Overall survival in patients with hepatocellular carcinoma

SECONDARY OUTCOMES:
progression-free survival | 3 years
  progression-free survival in patients with hepatocellular carcinoma
predictors of response to treatment | 3 years
  predictors of response to Atézolizumab and Bevacizumab
treatment tolerance | 3 years
  treatment tolerance to Atézolizumab and Bevacizumab

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Caen, Caen, France/Normandie, France